CLINICAL TRIAL: NCT06500312
Title: Assessment the Association of Imaging and Tumor Microenvironment in Lung Cancer With Radiogenomics
Brief Title: Decoding the Association of Imaging and Tumor Microenvironment in Lung Cancer Using Radiogenomic Approach（Radiogenomics-Lung）
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 0482
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is the prospective, observational cohort study (Radiogenomics-Lung), which aims to explore the relationship between the imaging information of lung cancer patients, tumor microenvironment and the prognosis of lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were treated for lung cancer in Wuhan Union Hospital from July 2024 to July 2027;
2. Aged > 18 years old;
3. At least one chest CT scan before treatment;
4. Tissue biopsy pathological examination confirmed the diagnosis of the above tumors.

Exclusion Criteria:

1. Poor image quality;
2. Incomplete clinical data or loss of follow-up;
3. Presence of another primary malignancy other than lung cancer;
4. Unclear pathological diagnosis。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were treated for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2027-07-02 (Estimated)

PRIMARY OUTCOMES:
Correlation analysis of sequencing results and body composition | 0.5 year
  Conducting correlation analysis between body composition and results of multi-omics sequencing
Correlation analysis of sequencing results and tumor radiomic features | 0.5 year
  Conducting correlation analysis between radiomic features and results of multi-omics sequencing

SECONDARY OUTCOMES:
Constructing tumor microenvironment prediction model | 2 years
  Constructing radiomic model to predict tumor microenvironment. The indicator is the area under the curve (AUC) of the prediction model
Constructing a multi-dimensional prognostic prediction model | 3 years
  A high-dimensional model was constructed to predict the prognosis of patients through multi-omics sequencing data, body composition, and tumor radiomic features. The indicator is the area under the curve (AUC) of the prediction model.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China